CLINICAL TRIAL: NCT01089114
Title: Cardiovascular Radiologic and Metabolic Assessment in HIV: An Investigation of Pathophysiology
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100080; 10-I-0080
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2015-08-07

CONDITIONS: HIV; Cardiovascular Disease
Keywords: Cardiac Imaging; MR Spectroscopy; HIV; Lipid Metabolism; HIV Infection; Cardiovascular Disease; HIV Infections
MeSH Terms: conditions — Cardiovascular Diseases; HIV Infections

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Antiretroviral therapy has increased the lifespan of people with human immunodeficiency virus (HIV), but recent research suggests that people with HIV also have an increased risk of developing cardiovascular disease. To better understand the prevalence and effects of heart disease in people with HIV, researchers are interested in comparing heart imaging and metabolism studies to see if there are differences between HIV-positive and HIV-negative people.

Objectives:

- To study metabolism and heart function in people with HIV compared with healthy HIV-negative volunteers.

Eligibility:

- Individuals at least 18 years of age who either have been diagnosed with HIV or are healthy HIV-negative volunteers.

Design:

* Participants will be evaluated with a physical exam, detailed medical history, and routine blood and urine tests including HIV testing.
* Participants will have the following imaging scans:
* Cardiac magnetic resonance imaging (MRI) to study the health of the heart and blood vessels
* Magnetic resonance spectroscopy (MRS) of the heart, liver, and skeletal muscle
* Cardiac computerized tomography (CT) scan to measure calcium levels in the heart and nearby arteries
* Dual-energy x-ray absorptiometry (DEXA) scan to measure body fat and muscle mass.
* Stable isotope infusion to evaluate how the body processes fat (which will require an overnight stay before the test)
* Participants will also have blood tests, an echocardiogram, and an electrocardiogram to evaluate heart function.

DETAILED DESCRIPTION:
HIV is now a chronic infection as patients with access to antiretroviral therapy have significantly improved life expectancies. Patients with HIV also have an increased risk of cardiovascular disease. Thus, cardiovascular disease is an important potential co-morbidity for patients living with HIV. The current proposal will perform a detailed cardiovascular assessment using state-of-the-art imaging techniques to evaluate intramyocardial lipid as well as coronary artery disease and myocardial function in a cohort of 100 HIV infected patients and 30 healthy volunteers as controls. This is an early exploratory cross-sectional study designed to both assess the burden of disease and apply novel techniques in this unique population.

ELIGIBILITY:
* HIV-Infected Participants Criteria:

INCLUSION CRITERIA:

1. Age 18 years or greater
2. Documented HIV infection
3. Willingness to have stored samples

EXCLUSION CRITERIA:

1. Subject is deemed unable to comply with requirements of study participation.
2. Subjects with contraindication to MRI scanning. These contraindications include but are not limited to the following devices or conditions:

   * Implanted cardiac pacemaker or defibrillator
   * Cochlear implants
   * Ocular foreign body (e.g. metal shavings)
   * Embedded shrapnel fragments
   * Central nervous system aneurysm clips
   * Implanted neural stimulator
   * Medical infusion pumps
   * Any implanted device that is incompatible with MRI.
3. Subjects requiring sedation for MRI studies.
4. Subjects with a condition precluding entry into scanner and acquisition of scans (e.g. morbid obesity, claustrophobia, back pain, motion disorders).
5. Women who are lactating, pregnant, or actively seeking to become pregnant.
6. History of severe allergic reaction to gadolinium contrast agents despite the use of premedication with an anti-histaminic and cortisone.
7. Estimated glomerular filtration rate (eGFR) <60 cc/min/1.73m(2).
8. Creatinine value >3.0 mg/dl

For Coronary CTA with Iodine-Based Contrast*:

1. Contraindication to the use of CT contrast agents:

   * Creatinine value >1.4 mg/dl or eGFR <60 cc/min/1.73m(2).
   * History of multiple myeloma
   * Use of metformin-containing products less than 24 hrs prior to contrast administration
   * History of significant allergic reaction to CT contrast agents
2. Subjects with contraindication precluding the use of beta blockers necessary to perform the coronary CTA. These include:

   * Clinically significant asthma
   * Active bronchospasm
   * Moderate or severe chronic obstructive pulmonary disease (COPD)
   * 2nd or 3rd degree AV block
   * Decompensated cardiac failure
   * Allergy to beta blockers
   * Systolic blood pressure <100 mm Hg
3. Guidelines for use of beta blocker is outlined in Appendix 1.

   * Participants who are eligible for MRI but who are not eligible for cardiac CT scan will be allowed to participate in the non-CT portion of the study.

Healthy Control Criteria:

INCLUSION CRITERIA:

1. Age 18 years or greater
2. Willingness to have stored samples

EXCLUSION CRITERIA:

All of the exclusion criteria for HIV-infected participants listed above apply to healthy controls. In addition, the following exclusion criteria will also be applied to healthy controls:

1. Clinically significant, systemic illness (serious infections or significant cardiac, pulmonary, hepatic, or other organ dysfunction) which in the judgment of the investigators would compromise the patient s ability to tolerate this study.
2. History of or current known cardiovascular disease.
3. HIV infection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-03-08; Study Completion 2015-08-07

PRIMARY OUTCOMES:
Intramyocardial triglyceride

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Hadigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] DAD Study Group; Friis-Moller N, Reiss P, Sabin CA, Weber R, Monforte Ad, El-Sadr W, Thiebaut R, De Wit S, Kirk O, Fontas E, Law MG, Phillips A, Lundgren JD. Class of antiretroviral drugs and the risk of myocardial infarction. N Engl J Med. 2007 Apr 26;356(17):1723-35. doi: 10.1056/NEJMoa062744. PMID 17460226
- [Background] Triant VA, Lee H, Hadigan C, Grinspoon SK. Increased acute myocardial infarction rates and cardiovascular risk factors among patients with human immunodeficiency virus disease. J Clin Endocrinol Metab. 2007 Jul;92(7):2506-12. doi: 10.1210/jc.2006-2190. Epub 2007 Apr 24. PMID 17456578
- [Background] Hsue PY, Hunt PW, Ho JE, Farah HH, Schnell A, Hoh R, Martin JN, Deeks SG, Bolger AF. Impact of HIV infection on diastolic function and left ventricular mass. Circ Heart Fail. 2010 Jan;3(1):132-9. doi: 10.1161/CIRCHEARTFAILURE.109.854943. Epub 2009 Nov 20. PMID 19933410